CLINICAL TRIAL: NCT00287261
Title: A Prospective Multicentre Phase II Trial of Zoledronic Acid in Patients With Myelofibrosis With Myeloid Metaplasia (MMM)
Brief Title: A Trial of Zoledronic Acid in Patients With Myelofibrosis With Myeloid Metaplasia (MMM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Hans Wildiers, adjuvnt head of clinic, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446G2422
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Myelofibrosis; Myeloid Metaplasia
Keywords: myelofibrosis; D009191
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- zometa (Experimental): 3-weekly infusion of zometa (zoledronic acid) 4 mg
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — 4 mg IV every 3 weeks for 36 weeks

SUMMARY:
In this trial, the question is addressed if zoledronic acid (Zometa, Novartis Pharma)could be of clinical benefit for patients with myelofibrosis and myeloid metaplasia (MMM).

DETAILED DESCRIPTION:
This is a prospective, multicentre phase II study in adult patients with documented MMM and requiring therapy for their disease. Patients will be treated every 3 weeks with 4 mg zoledronic acid (Zometa), administered by a 15 min. intravenous infusion. Study duration is 36 weeks (12 infusions). After the study it is recommended to continue treatment until disease progression, or the occurrence of unacceptable treatment-related toxicity.

Objectives of the trial are:

Primary objectives: the effect of monthly infusion of zoledronic acid 4 mg on:

hemoglobin level, spleen size

Secondary objectives the effect of monthly infusion of zoledronic acid 4 mg on: red blood cell transfusion need performance status constitutional symptoms leukocyte count thrombocyte count bone marrow fibrosis serum LDH

ELIGIBILITY:
Inclusion Criteria:

male or female and at least 18 years-of-age histologically confirmed diagnosis of myelofibrosis with myeloid metaplasia (MMM). This includes patients with agnogenic myeloid metaplasia (also known as idiopathic myelofibrosis) and patients with a preceding history of polycythemia vera or essential thrombocytemia (also known as post-polycytemic myelofibrosis). (see Appendix A) patients with low, intermediate and high risk disease categories (following the Dupriez score) may be included presence of measurable, clinically relevant disease manifestations (especially for low risk patients) ECOG performance status of 0, 1 or 2 life expectancy of at least 3 months Women of childbearing potential must use a medically acceptable form of contraception during the study and must have a negative urine or serum pregnancy test within 7 days of randomization written informed consent

Exclusion Criteria:

diseases associated with secondary myelofibrosis, such as metastatic carcinoma, lymphoma, myelodysplasia, hairy cell leukemia, mast cell disease, acute leukemia (including M7 disease or acute panmyelosis with myelofibrosis) presence of the chromosomal translocation t(9:22) or molecular BCR/ABL rearrangement as detected by RT-PCR in bone marrow or peripheral blood any anti-myelofibrosis drug therapy during the last 4 weeks. This includes chemotherapy, androgens, steroids, thalidomide, hematopoietic growth factors or any other investigational drug patients that have received bisphosphonates in the previous 3 months known allergy or intolerance to bisphosphonates abnormal renal function as evidenced by: a calculated creatinine clearance < 30 ml/min (creatinine clearance (CrCl) is calculated using the Cockcroft and Gault formula) (see Appendix F) corrected serum calcium < 8.0 mg/dL . Corrected serum calcium (mg/dl) = measured calcium (mg/dl) + 0.8*[4 - patient serum albumin (g/dl)] patients with nonmalignant conditions which would confound the evaluation of the primary endpoint, impair tolerance of therapy, or prevent compliance to the protocol, including: uncontrolled infections uncontrolled type 2 Diabetes Mellitus diseases with influence on bone metabolism such as Paget's disease or uncontrolled thyroid or parathyroid dysfunction cardiovascular, renal, hepatic, pulmonary and neurologic/psychiatric diseases which would prevent prolonged follow-up current active dental problems including infection of the teeth or jawbone (maxilla or mandibula); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw, of exposed bone in the mouth, or of slow healing after dental procedures recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants) patients with a history of non-compliance to medical regimens and patients who are considered potentially unreliable and/or not cooperative patients treated with any systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days pregnant or breast feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
effect of monthly zoledronic acid infusion on hemoglobin level and spleen size | 36 weeks

SECONDARY OUTCOMES:
red blood cell transfusion need | 36 weeks
performance status | 36 weeks
constitutional symptoms | 36 weeks
leukocyte count | 36 weeks
thrombocyte count | 36 weeks
serum LDH | 36 weeks
bone marrow histology | 36 weeks
safety of zometa infusions | until progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delforge, MD, PhD, Principal Investigator — University Hospital Leuven, Belgium
Locations (6):
- Cancer Care Services, Brisbane, Queensland, Australia
- University Hospital Leuven, Leuven, Belgium
- Hopital Avicenne and Paris 13 University, Bobigny, France
- Medizinische Klinik Kiel, Kiel, Germany
- RAMBAM Medical Center and Technion, Haifa, Israel
- Hospital Rafael éndez, Murcia, Lorca, Spain